CLINICAL TRIAL: NCT02274103
Title: Improving Health Through SkypeTM: Family-Based Intervention for Teens With Poorly Controlled Diabetes
Brief Title: Skype for Youth With Poorly Controlled Diabetes
Acronym: SKYPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Michael A. Harris, PhD, Professor, Pediatrics, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6000
Record Dates: First submitted 2014-10-21; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinic (Active Comparator): BFST delivered to youth with poorly controlled diabetes and their families in the clinic, face-to-face.
  Interventions: Behavioral: BFST
- Skype (Active Comparator): BFST delivered to youth with poorly controlled diabetes and their families using Skype.
  Interventions: Behavioral: BFST

INTERVENTIONS:
Behavioral: BFST — Family-based skills training.

SUMMARY:
Compared family-based skills training (aka, Behavioral Family Systems Therapy) to youth with poorly controlled type 1 diabetes and their parents either face-to-face or over SkypeTM. Examined the differential impact on the youth's adherence to the diabetes medical regimen and the youth's blood sugar control.

ELIGIBILITY:
Inclusion Criteria:

* Youth between the ages of 12 and 18 with type 1 diabetes characterized by an HbA1c value great than 9%
* Caregivers willing to participate
* Family members reading English at 5th grade level
* Willing to be randomized.

Exclusion Criteria:

* Youth with intellectual disability
* Parent or youth who doesn't speak English

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from Baseline to 3 months and from 3 months to 6 months
  HbA1c values for both intervention groups improved from baseline to 3 months and from 3 months to 6 months.

SECONDARY OUTCOMES:
Adherence to diabetes treatment using the Diabetes Self Management Profile (DSMP) (Harris et al, 2001). | Change from Baseline to 3 months and from 3 months to 6 months
  DSMP scores for both intervention groups improved from baseline to 3 months and from 3 months to 6 months.

REFERENCES:
- [Derived] Duke DC, Wagner DV, Ulrich J, Freeman KA, Harris MA. Videoconferencing for Teens With Diabetes: Family Matters. J Diabetes Sci Technol. 2016 Jun 28;10(4):816-23. doi: 10.1177/1932296816642577. Print 2016 Jul. PMID 27075708
- [Derived] Harris MA, Freeman KA, Duke DC. Seeing Is Believing: Using Skype to Improve Diabetes Outcomes in Youth. Diabetes Care. 2015 Aug;38(8):1427-34. doi: 10.2337/dc14-2469. Epub 2015 Jun 1. PMID 26033508
- [Derived] Riley AR, Duke DC, Freeman KA, Hood KK, Harris MA. Depressive Symptoms in a Trial Behavioral Family Systems Therapy for Diabetes: A Post Hoc Analysis of Change. Diabetes Care. 2015 Aug;38(8):1435-40. doi: 10.2337/dc14-2519. Epub 2015 May 26. PMID 26015558